CLINICAL TRIAL: NCT01430572
Title: Phase I Combination of Pazopanib and Everolimus in PI3KCA Mutation Positive/PTEN Loss Patients With Advanced Solid Tumors Refractory to Standard Therapy
Brief Title: Pazopanib and Everolimus in PI3KCA Mutation Positive/PTEN Loss Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0322; NCCN-GSKP05 (Other: NCCN); NCI-2011-03040 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Advanced Cancers; Solid Tumors
Keywords: Advanced Cancers; Solid Tumors; PI3KCA Mutation Positive/PTEN; Refractory to standard therapy; Relapsed after standard therapy; Pazopanib; GW786034; Everolimus; Afinitor; RAD001
MeSH Terms: interventions — pazopanib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pazopanib + Everolimus (Experimental): Pazopanib 200 mg and Everolimus 5.0 mg oral dosing every other day (except for lead in 5 days of Cycle 1 where both drugs administered daily).
  Interventions: Drug: Pazopanib; Drug: Everolimus

INTERVENTIONS:
Drug: Pazopanib — Starting Dose: 200 mg by mouth on Days 1 - 5 of Cycle 1 only. On Day 6 and every cycle-day with an even number, only pazopanib administered.
  Other Names: GW786034
Drug: Everolimus — Starting dose: 5.0 mg by mouth on Days 1 - 5 of Cycle 1. On Day 7 and every cycle-day with an odd number, only everolimus will be administered.
  Dose Expansion Phase: Maximum tolerated dose (MTD) from lead in phase.
  Other Names: Afinitor; RAD001

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of Votrient (pazopanib) and Afinitor (everolimus) that can be given to patients with advanced cancer. The safety of these drugs will also be studied.

Pazopanib is designed to block different receptors in the cancer cells that ultimately are responsible for the growth of the tumor and its blood vessels.

Everolimus is designed to block a protein called mTOR inside the cancer cells, which is also involved in cancer growth.

DETAILED DESCRIPTION:
Study Groups:

Dose Escalation:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of the combination of pazopanib and everolimus based on when you joined this study. Up to 8 dose levels of pazopanib and everolimus will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of pazopanib and everolimus is found.

Expansion:

Once the highest tolerable dose of pazopanib and everolimus is found, up to 14 more participants may be enrolled to further study the safety of the drugs at that dose and the efficacy of the drugs in a certain tumor group.

Study Drug Administration:

Each study cycle is 28 days.

Pazopanib and everolimus are taken by mouth on an empty stomach (1 hour before meals or 2 hours after meals).

On Days 1-5 of Cycle 1 only, you will take pazopanib and everolimus together. First take pazopanib and then take everolimus.

After those first 5 days, you will take pazopanib and everolimus every other day separately. Starting Day 6 of Cycle 1, pazopanib will be taken every even day (6, 8, 10, and so on) . Everolimus will be taken every odd day (7, 9, 11, and so on).

Beginning with Cycle 2, you will take pazopanib every even day (2, 4, 6, and on so) and everolimus every odd day (3, 5, 7, and so on).

Study Visits:

At each study visit, you will be asked what about any drugs or herbal supplements that you may be taking and if you have had any side effects.

On Day 1 of Cycle 1:

* Your medical history will be recorded if it has been more than 3 days since screening.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will have an ECG.
* Blood (about 2 teaspoons) and urine will be collected for routine tests and hepatitis screening.

On Days 8, 15, and 22 of Cycle 1:

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.

On Day 1 of Cycles 2 and beyond:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* You will have an ECG.

On Day 15 of Cycle 2:

° Blood (about 2 teaspoons) will be collected for routine tests.

Every 8 weeks:

* You will have a CT scan, x-ray, MRI scan, and/or PET scan to check the status of the disease.
* Blood (about 1 teaspoon) may be drawn for tumor marker testing.
* If you are able to become pregnant, you will have a blood (about ½ teaspoon) or urine pregnancy test.

PK testing:

At least 6 participants in the expansion part of the study will have blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing. The study staff will tell you if you will have this testing. PK testing measures the amount of study drug in the body at different time points.

* On Day 5 of Cycle 1 and Days 1 and 2 of Cycle 2, blood will be drawn before and 8 more times up to 10 hours after taking the study drugs.
* On Day 2 of Cycle 2, blood will be drawn 1 more time for PK testing after 24 hours of taking everolimus. If you could not have the 10 hour draw the day before, this will be drawn at this day.
* On Day 6 of Cycle 1 and Day 3 of Cycle 2, blood will be drawn 1 time for PK testing after 24 hours of taking pazopanib. If you could not have the 10 hour draw the day before, this will be drawn at this day.
* Blood will be drawn 1 time at the end-of-dosing visit.

Length of Study:

You may continue taking the study drugs for as long as you are benefitting. You will be taken off study early if the disease gets worse, intolerable side effects occur, you develop new health problems, or your doctor thinks that it is no longer in your best interest to receive the study drug.

End-of-Dosing Visit:

Within 4 weeks after your last dose of study drugs:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.

This is an investigational study. Pazopanib is FDA approved and commercially available for the treatment of advanced renal cancer and certain types of advanced soft tissue sarcoma but has not been approved for use in other cancer types. Everolimus is FDA approved and commercially available for the prevention of kidney transplant rejection, to treat advanced renal cancer, and to treat subependymal giant cell astrocytoma associated with tuberous sclerosis.

The combination of pazopanib and everolimus to treat advanced cancer is investigational.

Up to 62 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up.
2. Patients with advanced or metastatic solid tumors that are refractory to standard therapy, relapsed after standard therapy, or who have no standard therapy available that improves survival by at least three months.
3. Patients must have been off previous chemotherapy or radiotherapy for two weeks prior to start of treatment. For biologic/targeted therapies, patients must be >/= five half-lives or >/= 2 weeks from the last treatment dose, whichever comes first. Patients may have received palliative localized radiation immediately before (or during) treatment provided radiation is not delivered to the single target lesion available.
4. ECOG performance status </= 2.
5. Abnormal organ function is permitted. However, patients must meet the following criteria: neutrophil count >/= 1.5 x 10*9/L; platelets >/= 100 x 10*9/L; creatinine </= 1.5 X upper limit of normal (ULN); T. bilirubin </= 1.5 X ULN; AST(SGOT) and/or ALT(SGPT) </= 2.5 X ULN, UPC < 1.
6. Women of child-bearing potential MUST have a negative serum or urine HCG test within 14 days of first dose. Sexually active patients must agree to use contraception for the duration of study participation: women, 2 weeks before the first treatment dose and for 28 days after the last dose; and men, from the first treatment dose and for 28 days after the last dose of treatment. For the purpose of this protocol women of child-bearing potential are defined as: a female able to have children that has not been surgically sterilized or that has not been without menses for 12 consecutive months.
7. Patients must be >/=16 years of age.
8. Fresh blood samples must be provided for all subjects for biomarker analysis before treatment with investigational product.
9. Patients must have evaluable disease by RECIST criteria.
10. For the dose expansion cohort patients will have to have any kind of genomic alteration in either PI3K and/or PTEN of their tumor.

Exclusion Criteria:

1. Central nervous system (CNS) metastases at baseline, with the exception of those subjects who have previously-treated CNS metastases (surgery +/- radiotherapy, radiosurgery, or gamma knife) and who meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or enzyme-inducing anti-convulsants in prior 2 weeks.
2. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:Active peptic ulcer disease; Known intraluminal metastatic lesion/s with risk of bleeding; Inflammatory bowel disease (e.g. ulcerative colitis, Chrohn's disease),or other gastrointestinal conditions with increased risk of perforation; History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior beginning study treatment.
3. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to; Malabsorption syndrome; Major resection of the stomach or small bowel
4. Corrected QT (QTc) > 480 msecs.
5. History of any one or more of the following cardiovascular conditions within the past 6 months:Cerebrovascular accident, Myocardial infarction, Unstable angina , Cardiac angioplasty or stenting, Coronary artery bypass graft surgery, Class III or IV heart failure, as defined by the New York Heart Association (NYHA), Untreated pulmonary embolism (PE) or deep venous thrombosis (DVT). Note: subjects with recent PE or DVT who have been therapeutically coagulated for at least 6 weeks are eligible.
6. Uncontrolled systemic vascular hypertension (systolic blood pressure >/= 140 mmHg, diastolic blood pressure >/= 90 mmHg). Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals. At least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement. These three values should be averaged to obtain the mean diastolic BP and mean systolic BP. The mean SBP/DBP ration must be < 140/90.
7. Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
8. Evidence of active bleeding or bleeding diathesis.
9. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage. Note: Lesions infiltrating major pulmonary vessels (contiguous tumor and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating (abutting) the vessels is acceptable (CT with contrast is strongly recommended to evaluate such lesions). Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed. Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed.
10. Recent hemoptysis (>/= ½ teaspoon of red blood within 8 weeks before first dose of study drug).
11. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
12. Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment.
13. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.
14. Prior malignancy Note: Subjects who have had another malignancy and have been disease-free for 2 years, and/or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-10-07 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Pazopanib and Everolimus | 28 days
  MTD defined as highest dose studied in which the incidence of Dose Limiting Toxicity (DLT) was less than 33%, with no more than 1 of 6 evaluable participants had a DLT using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Response.of Pazopanib and Everolimus | 4 months
  Response evaluated using following criteria: Stable disease for more than or equal to 4 months.
Response.of Pazopanib and Everolimus | 4 months
  Response evaluated using following criteria: Decrease in measurable tumor (target lesions) by more than or equal to 20% by RECIST criteria.
Response.of Pazopanib and Everolimus | 4 months
  Response evaluated using following criteria: Decrease in tumor markers by more than or equal to 25% (for example, a >/= 25% decrease in PSA for patients with prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org